CLINICAL TRIAL: NCT04581941
Title: Deep Brain Stimulation Effects in Essential Tremor: Time Course of Electrophysiological Changes in Treatment
Brief Title: Deep Brain Stimulation Effects in Essential Tremor
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202002623
Record Dates: First submitted 2020-10-06; First posted 2020-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with essential tremor: Patients with essential tremor who have clinically been deemed candidates for DBS (Deep Brain Stimulation) surgery. Deep brain stimulation is an FDA approved therapy that involves surgical implantation of electrodes in deep brain targets and an implantable pulse generator delivers electrical pulses. This intervention is not part of the study. The investigators are going to recruit patients who receive the Medtronic Percept device, which allows for brain signal recordings (this feature is FDA approved). The investigators will be conducting an observational study using this device to collect data that the subjects receive as standard of care.

SUMMARY:
Deep Brain Stimulation (DBS) is an effective therapy for patients with medically refractory essential tremor. However, DBS programming is not standardized and multiple clinic visits are frequently required to adequately control symptoms. The investigators aim to longitudinally record brain signals from patients using a novel neurostimulator that can record brain signals. The investigators will correlate brain signals to clinical severity scores to identify pathological rhythms in the absence of DBS, and we will study the effects of DBS on these signals in order to guide clinical programming.

DETAILED DESCRIPTION:
The development of newer technologies has allowed clinicians and researchers to better understand pathophysiological underpinnings of different disorders managed with neuromodulation. The is now the ability to stream brain signals from a newly FDA approved device, the Medtronic Percept. The investigators will study the longitudinal effects of DBS on the brain signals that are found to correlate with tremor severity as measured with wireless wearable sensors.

ELIGIBILITY:
Inclusion Criteria

* Patient gives an informed consent.
* Patient is over 21 years of age.
* Having a diagnosis of a essential tremor confirmed by a trained movement disorders neurologist;
* Having failed or not tolerated conventional medical management, at the discretion of the neurologist managing the patient;

Exclusion Criteria

* Having alternative diagnoses to essential tremor;
* Having comorbid neurodegenerative disorders that may affect mobility or cognition (e.g. comorbid Parkinson's disease or dystonia);
* Having sequelae of prior brain insult (e.g. prior stroke or brain tumor);
* History of prior resective brain surgery (e.g. tumor resection);
* Not being a DBS candidate;
* Receiving unilateral implants
* Having a higher surgical risk that precludes patient from having standard intraoperative mapping.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with essential tremor, who have been cleared for DBS surgery.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Fahn- Tolosa- Marin Tremor Rating Scale | 6 months
  A clinical scale of tremor severity (0-4, 0:no symptoms, 4:extreme)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States